CLINICAL TRIAL: NCT04838184
Title: Prospective Clinical Study of Straumann Roxolid®/SLactive® Short Implants in Edentulous Mandible
Brief Title: Short Implants in Edentulous Mandible
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Straumann AG (Unknown)
Responsible Party: Sponsor
Other Study IDs: PV_4805
Record Dates: First submitted 2021-03-18; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Tooth Loss; Edentulous Jaw
MeSH Terms: conditions — Tooth Loss; Jaw, Edentulous | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental patients: Patients with an edentulous mandible who are demanding and receiving an implant-supported fixed dental prosthesis in the mandible
  Interventions: Device: Dental Implants (Straumann Roxolid® / SLActive®)

INTERVENTIONS:
Device: Dental Implants (Straumann Roxolid® / SLActive®) — In this study the 4 mm implants will be inserted in the area surrounding 36/46. The implant diameters will be defined based on the patient's situation.
  In the interforaminal region, two implants of conventional length with a minimum of 10 mm will be inserted. The implant diameter and the length will be defined based on the patient's situation.

SUMMARY:
Main aim of this study was to assess survival rates of short implants with a length of 4 mm in the edentulous mandible after 1, 3, and 5 years.

DETAILED DESCRIPTION:
It is hypothesized that survival rates after 1, 3, and 5 years of Straumann Roxolid® / SLActive® 4 mm short implants do not differ from values of Straumann SLActive implants with more than 4 mm length in the same clinical situation.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* Age: 18 to 70
* Edentulous mandible with reduced bone level in the posterior region (> 5 mm and < 8 mm above nerve conduit)
* Physical and mental condition that allow surgery and a 5-year follow-up period to be carried out without foreseeable problems
* Obtained informed consent from the patient

Specific criteria:

* Limited vertical space for implant placement, where conventional implants with lengths of more than 4 mm cannot be used
* Tooth loss or extraction at least 8 weeks before implant surgery
* Healthy implantation site
* Favorable and stable occlusal relationship
* Complete denture in the mandible. If no denture available, an interims prosthesis will be fitted
* Natural full dentition or sufficient complete or partial dentures in the maxilla

Exclusion Criteria:

General criteria:

* Any conditions or circumstances which would interfere with the requirements for oral surgery
* Allergy to any metallic implant component
* Acute, untreated periodontitis
* Previous oro-maxillo-facial radiotherapy
* Any disorders in the planned implant area such as previous tumors or chronic bone disease (e.g., rheumatoid disease)
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc.)
* Alcohol or drug abuse
* Heavy smoking (>10 cigarettes/day)
* Uncontrolled diabetes
* Severe bruxism or other destructive oral habits
* Pregnant or lactating women

Specific criteria:

* Need for a major bone regeneration technique
* Infections in adjacent tissue of the planned implantation site.
* Bleeding on probing (BOP) and plaque index (PI) higher 25%
* Insufficient bone volume in the posterior region for placing a Straumann Roxolid® / SLActive® 4mm short implant and in the interforaminal region for placing a Straumann Roxolid® / SLActive® implant with a minimum length of 10 mm determined by radiographic analysis (OPG)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental patients of university-based prosthodontic department (primary, secondary, and tertiary care clinic)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-04-19 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 years
  Survival of implants and suprastructure. Measure: survival rates

SECONDARY OUTCOMES:
Implant stability | 3 months
  Within-subject comparison of primary (at implant placement) and secondary (at implant exposure) stability of short versus regular length implants.
  Measure / device: Resonance Frequency Analysis (RFA)
Success | 5 years
  Success of implants and suprastructure. Measure: success rates
  * Biological success:
    * No detectable clinical mobility (hand testing)
    * No radiolucency surrounding the total surface of the implant
    * No persistent pain refractory to medical therapy
    * No recurrent peri-implant infection
      * Peri-implant infection: peri-implant Probing Depth (PD), Plaque Index (Pl), and Bleeding on Probing (BoP)
      * Bone loss: standardized intra-oral radiography with long-cone parallel technique
  * Technical success:
    * No screw loosening
    * No fracture of metal base
    * No fracture of veneering material
Oral health-related quality of life | 5 years
  Oral health-related quality of life (OHRQoL). Measure: questionnaire
  - 49-item Oral Health Impact Profile (OHIP) with a 5-point ordinal rating scale (possible range of summary scores: 0-196 with higher scores indicating more impairment)
Patient satisfaction | 5 years
  Patient satisfaction. Measure: questionnaire
  - Visual analogue scales (VAS) on ease of cleaning, speech, comfort, esthetic, stability, chewing ability, masticatory function, and oral health (possible range of scores: 0-10 for each item with higher scores indicating more satisfaction)

IPD SHARING:
Plan to Share IPD: No